CLINICAL TRIAL: NCT06035133
Title: One Arm Exploratory Trial of Efficacy and Safety of TNT Plus Mode With Neoadjuvant Radiotherapy in the Treatment of Locally Advanced Medium-low Rectal Cancer
Brief Title: Treatment of Low Locally Advanced Rectal Cancer With Radiotherapy Removal TNT Plus Neoadjuvant Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202108-27
Record Dates: First submitted 2022-12-22; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab; Bevacizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy removal TNT plus group (Experimental): Six induction chemotherapy rounds of the CapeOX regimen were administered. RAS, BRAF, and MSI were found when the first patients were examined. Patients were given CapeOX + cetuximab for RAS wild-type patients, CapeOX + bevacizumab for RAS mutant patients, and CapeOX + cetuximab for MSI-H patients. The CapeOX regimen: Oxaliplatin 130 mg/m2, intravenous injection, day 1; capecitabine 1000 mg/m2, oral, twice daily, days 1 through 14; once every 3 weeks. A surgical procedure was carried out two weeks after consolidation chemotherapy ended.
  Interventions: Drug: CapeOX + cetuximab; Drug: CapeOX + bevacizumab; Radiation: radiotherapy

INTERVENTIONS:
Drug: CapeOX + cetuximab — CapeOX + cetuximab for RAS wild-type patients and CapeOX + cetuximab for MSI-H patients. The CapeOX regimen: Oxaliplatin 130 mg/m2, intravenous injection, day 1; capecitabine 1000 mg/m2, oral, twice daily, days 1 through 14; once every 3 weeks.
Drug: CapeOX + bevacizumab — CapeOX + bevacizumab for RAS mutant patients. The CapeOX regimen: Oxaliplatin 130 mg/m2, intravenous injection, day 1; capecitabine 1000 mg/m2, oral, twice daily, days 1 through 14; once every 3 weeks.
Radiation: radiotherapy — radiotherapy

SUMMARY:
(1) To evaluate the oncological effects of Treatment of low locally advanced rectal cancer with radiotherapy removal TNT plus neoadjuvant therapy TNT plus mode on TRG, Anal sphincter preservation surgery rate / rectal preservation surgery rate, cCR rate, pCR rate and other oncological effects in patients with middle and low LARC; (2) Evaluate the R0 resection rate, LARS score, urination function and sexual function score, local recurrence rate, and 3-year DFS and OS of Treatment of low locally advanced rectal cancer with radiotherapy removal TNT plus neoadjuvant therapy TNT plus mode, resolve the current dispute about the Treatment of low locally advanced rectal cancer with radiotherapy removal TNT plus neoadjuvant therapy TNT treatment mode of LARC, provide a new mode for LARC treatment, and hopefully rewrite the diagnosis and treatment guidelines for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70;
* Histologically confirmed adenocarcinoma of rectum;
* The distance from the lower edge of the tumor to the anus is ≤ 10cm;
* ECOG score ≤ 1;
* Have not received any anti-tumor treatment before;
* Preoperative abdominal enhanced CT or MRI showed cT4, cN0-2; M0 chest and abdomen CT showed no obvious metastasis. (Note: PET-CT is recommended when small nodules can not be identified by liver or lung CT, and can still be included in the group when considering the possibility of metastasis)
* Hematological indicators and liver and kidney function within 7 days are within the normal range;
* Sign the informed consent form and be able to follow the research and /or follow-up procedures.

Exclusion Criteria:

* Have serious basic diseases, such as heart disease, renal failure, severe liver failure or liver failure, coagulation dysfunction, etc; Postoperative recurrence of colorectal cancer;
* The patient had a history of malignant tumor within 5 years;
* Pregnant or lactating women;
* The patient has a history of adjuvant radiotherapy for other system diseases, and surgical contraindications, so it is not suitable for surgery;
* The patient has had radiotherapy and chemotherapy records before this visit;
* Distant metastasis was found during operation;
* Patients with poor radiotherapy compliance and difficult cooperation;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-11-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
tumor regression grading, TRG | one month after surgery
  Reference resist 1.1 rating